CLINICAL TRIAL: NCT03894254
Title: Predictive Factors Associated With Impairment in Functional Autonomy in a Regional Real-life Cohort of Patients With Alzheimer's Disease or Related Disorders (ADRD)
Brief Title: Predictive Factors of Autonomy Loss in Real-life Cohort
Acronym: MEM-AURA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 69HCL18_0613
Record Dates: First submitted 2019-03-25; First posted 2019-03-28 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Memory Disorders
MeSH Terms: conditions — Memory Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with subjective cognitive complaint or neurocognitive (Experimental): : Real-life cohort patients with subjective cognitive complaint or neurocognitive disorders undergoing medical examination in memory centers, and for whom extensive evaluations will be performed for the study
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — This is study carried out in current practice. Patients are undergoing a medical examination in a memory center, with extensive and systematic evaluations for the study involving the following tests: IADL, DAD6, New AGGIR, NPI, and mini-Zarit) assessing the functions (autonomy, behavior and caregiver burden).

SUMMARY:
The Alzheimer's disease or related disorders (ADRD) are among the most disabling diseases because of their main features such as cognitive impairment, loss of functional autonomy and behavioural disorders. In absence of current curative treatment, the identification of the predictive risk factors of progression of the disease, evaluated through its main symptoms, represents a major stake of public health. The Investigators aim at developing a regional database, which includes the patient medical records on a prospective basis, in collaboration with the medical and administrative staff and with the University hospital computer science departments.

The main objective is to study the predictive factors associated with change in functional autonomy level, measured every 6 to 12 months in centres across Region Auvergne Rhone-Alpes in France.

The real-life study population will consist in about 5400 patients with ADRD. The inclusion period will be of 3 years, the length of follow-up of each patient will be of 10 years max for a total study length of 13 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older, undergoing a medical visit in a memory center or neuro-cognition service
* Patients living at home or in housing
* Patients with memory impairment, at all stage of the disease

Exclusion Criteria:

* Patients in institution
* Patients under legal protection
* Patients with a hearing or visual impairment, which prevents carrying out examinations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5400 (Estimated)
Dates: Start 2020-09-09 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2032-03-01 (Estimated)

PRIMARY OUTCOMES:
Functional autonomy level | from 6 months to 12 months interval
  The Lawton Instrumental Activities of Daily Living (IADL)
Functional autonomy level | from 6 months to 12 months interval
  The Disability Assessment of Dementia (DAD-6)
Functional autonomy level | from 6 months to 12 months interval
  The New-AGGIR (French national score for dependency assessment)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Krolak-Salmon, PhD, Principal Investigator — Centre Mémoire de Ressources et de Recherche
Locations (5):
- France (5):
  - Hôpital Dugoujon, Caluire-et-Cuire
  - Centre Hospitalier Lyon Sud, Lyon
  - Service de neuro-cognition et neuro-ophtalmologie du Groupement Hospitalier Est, Lyon
  - CHU Saint-Etienne, Saint-Etienne
  - Centre Mémoire de Ressources et de Recherche de Lyon, Villeurbanne

IPD SHARING:
Plan to Share IPD: No